CLINICAL TRIAL: NCT04955236
Title: Partial Scalp Block Versus Fentanyl Infusion in Patients Undergoing Posterior Fossa Surgery Under General Anesthesia. A Randomized Control Trial
Brief Title: Partial Scalp Block in Posterior Fossa Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rania Samir Fahmy, Assistant professor of Anesthesia, ICU and pain medicine, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MS-317-2020
Record Dates: First submitted 2021-07-04; First posted 2021-07-08 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Posterior Fossa Tumor
Keywords: Partial scalp block; Posterior fossa surgery; Greater occipital nerve; Lesser occipital nerve; Third occipital nerve; Fentanyl
MeSH Terms: conditions — Infratentorial Neoplasms | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial scalp block (Experimental): Bilateral block of the greater lesser and third occipital nerves using bupivacaine 0.25% with epinephrine 1:200,000
  Interventions: Drug: Partial scalp block
- Fentanyl group (Active Comparator): Fentanyl infusion will be administered till time of dural closure
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Partial scalp block — Partial scalp blocks will be performed bilaterally after assuming the prone position.The Greater occipital will be blocked by injecting 3ml of local anaesthetic at a point half way between the mastoid process the external occipital protuberance along the superior nuchal line, medial to the occipital artery. The Lesser occipital nerve will be blocked by injecting 3ml of local anaesthetic infiltration along the superior nuchal line, 2.5 cm lateral to the greater occipital nerve block. The greater occipital nerve block also will cover the third occipital nerve due to the close location of the two nerves.
  A placebo infusion (normal saline) will be administered at the same rate as fentanyl infusion in the active comparator arm(1 µg/kg/hr.).
  Other Names: N
  Arms: Partial scalp block
Drug: Fentanyl — 1µg/kg/hr. of intravenous fentanyl infusion will be administered. A syringe filled with 20 ml of normal saline will be prepared and 3 ml of normal saline will be injected at the same points of the partial scalp block previously described
  Other Names: F
  Arms: Fentanyl group

SUMMARY:
Pain in patients undergoing posterior fossa surgery is regarded as more intense when compared to pain in patients undergoing supratentorial cranial surgeries. It may result in a rise in blood pressure and heart rate leading to serious effects as increased intracranial pressure and intracranial hemorrhage. For a long time, the control of pain has been the role of opioids. However, the use of opioids is not devoid of side effects. Hence, combining other techniques as partial scalp block with general anesthesia may be beneficial in controlling hemodynamics and decreasing the amount of opioids used without sacrificing the good quality of analgesia and anesthesia.

DETAILED DESCRIPTION:
Pain in patients undergoing posterior fossa surgery is regarded as more intense when compared to pain in patients undergoing supratentorial cranial surgeries. The main cause has been attributed to the substantial muscle dissection and trauma in this area.

Opioids remain as the current gold standard drugs for operative pain relief. However, exposure to large doses leads to multiple side effects of varying significance, such as nausea, vomiting, dizziness, constipation, respiratory depression, hypoventilation and disorders of breathing during sleep. Therefore, strategies other than opioids are recommended without sacrificing proper and effective analgesia.

Considering the previously mentioned facts, supplementing general anesthesia with regional anesthesia has been considered and was found to improve intraoperative hemodynamics, surgical field and postoperative analgesia.

In neurosurgery, scalp blocks and local anesthetic infiltration are being used along with general anesthesia either preoperatively to decrease the hemodynamic response to head pinning and surgical incision or postoperatively before emergence from anesthesia to decrease postoperative pain and result in a better outcome.

The current study aims to compare between partial scalp block(greater,lesser and third occipital nerve blocks) on the one hand versus fentanyl infusion on the other hand as pain controlling measures reflected on intraoperative hemodynamics in patients undergoing posterior fossa surgery.

After approval of ethics research committee and obtaining informed written consents from the patient's first degree relatives, 40 patients will be randomly divided by computer designed lists and then concealed in closed serially numbered, opaque envelopes into 2 equal groups to receive either partial scalp block(greater,lesser and third occipital nerve blocks) or fentanyl infusion after induction of general anesthesia by a conventional method and assuming the prone position.

For group N (partial nerve block group): The scalp blocks will be performed bilaterally after assuming the prone position by an anesthesiologist who will not be a part of the study team nor will be involved in the proceeding data analysis or other parts of the study. The Greater occipital will be blocked by injecting 3ml of local anaesthetic at a point half way between the mastoid process the external occipital protuberance along the superior nuchal line, medial to the occipital artery. The Lesser occipital nerve will be blocked by injecting 3ml of local anaesthetic infiltration along the superior nuchal line, 2.5 cm lateral to the greater occipital nerve block. The greater occipital nerve block will also cover the third occipital nerve due to the close location of the two nerves (8).

To anesthetize the dura Lidocaine soaked gauzes will be used and applied for 10 minutes before dural incision.

A placebo infusion (normal saline) was administered at the same rate as fentanyl infusion (1 µg/kg/hr.).

For group F ( Fentanyl group):1µg/kg/hr. of intravenous fentanyl infusion will be administered. A syringe filled with 20 ml of normal saline will be prepared and 3 ml of normal saline will be injected at the same points of the partial scalp block previously mentioned. Both the syringe containing bupivacaine and adrenaline and the placebo syringe will be prepared by a blinded clinical pharmacist, who will not be a part of the study team nor will be involved in the proceeding data analysis or other parts of the study.

The primary outcome will be the systolic blood pressure at time of skin incision. the sample size was calculated using the medcalc software. Based on the study "Bupivacaine scalp nerve block: Hemodynamic response during craniotomy, intraoperative and post-operative analgesia" published in Asian biomedicine (2010).

The total sample size required was 36 participants to be randomly allocated between two groups to achieve a confidence level of 95%, power of study 80% with confidence interval of 1. The sample size was increased to 40 (20 per group) to guard against dropouts.

SPSS software will be used for data analysis. Categorical data will be expressed as frequencies and percentages and will be analyzed using chi-square test. Continuous data will be tested for normality by means of shapiro-wilk test and will be analyzed using unpaired t test, Mann Whitney test, and analysis of variance test (ANOVA) as appropriate. The numerical data will be presented as mean and standard deviation or median and interquartile range as appropriate. A P value less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Physical status ASA I and ASA ll.
* Males and females between the ages of 21 and 55.
* Patients undergoing posterior fossa Surgeries.
* Patients with GCS ≥14
* Patients undergoing operation in prone position

Exclusion Criteria:

* Patient refusal.
* Patients with a history of allergy to opioids or local anesthetics
* GCS (Glasgow coma score) ≤13 upon emergence from anesthesia.
* Patients who will need post-operative ventilation
* Patients who had previous craniotomies
* Patients with contraindication to regional anaesthesia e.g.: local sepsis,
* Patients with pre-existing peripheral neuropathies and coagulopathy.
* Patients who will develop intraoperative surgical complications
* Operations lasting more than 5 hours.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure at time of skin incision | During surgery, 1 min after skin incision
  Recording of the systolic blood pressure in mmhg at the time of skin incision

SECONDARY OUTCOMES:
Number of intraoperative fentanyl boluses | During surgery
  Total fentanyl boluses in micrograms which will be administered intraoperatively when heart rate and/or systolic arterial pressure values will exceed the baseline values by 25%
RASS score | One hour after the surgery
  Richmond agitation sedation score is a score used to describe the patients' level of alertness or agitation. It ranges from from -5 unarousable to +4 combative with 0 meaning alert and calm
Time for first rescue Analgesia | after the surgery
  First time when the patient starts to complain of pain after surgery and an analgesic is given
Number of heart beats per minute (Heart rate) | baseline, 5 min after the induction of anesthesia, 5 min after the scalp block, 1 min after skin incision, 1min after dural incision, at time of dural closure, 1 min after skin closure, at time of extubation.
  Number of heart beats per minute
Systolic blood pressure | baseline, 5 min after the induction of anesthesia, 5 min after the scalp block, 1 min after dural incision, at time of dural closure, 1 min after skin closure, at time of extubation.
  systolic blood pressure in mmhg
Mean arterial blood pressure | baseline, 5 min after the induction of anesthesia, 5 min after the scalp block, 1 min after skin incision, 1 min after dural incision, at time of dural closure, 1 min after skin closure, at time of extubation.
  Mean arterial blood pressure in mmhg
Diastolic blood pressure | baseline, 5 min after the induction of anesthesia, 5 min after the scalp block, 1 min after skin incision, 1 min after dural incision, at time of dural closure, 1 min after skin closure, at time of extubation.
  Diastolic blood pressure in mmhg
Intraoperative phentolamine consumption | throughout the operation
  the total amount of phentolamine in mg consumed intraoperatively
Intraoperative ephedrine consumption | throughout the operation
  the total amount of ephedrine in mg consumed intraoperatively
Time to extubation | At the end of the operation, the time from the discontinuation of inhalation agents till extubation
  It is the time between closure of inhalational anesthetic and extubation

CONTACTS AND LOCATIONS:
Overall Officials: Rania S Fahmy, Principal Investigator — Kasr Al Ainy, Faculty of medicine, Cairo university
Locations (1):
- Kasr El Aini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vadivelu N, Kai AM, Tran D, Kodumudi G, Legler A, Ayrian E. Options for perioperative pain management in neurosurgery. J Pain Res. 2016 Feb 10;9:37-47. doi: 10.2147/JPR.S85782. eCollection 2016. PMID 26929661
- [Background] Pinosky ML, Fishman RL, Reeves ST, Harvey SC, Patel S, Palesch Y, Dorman BH. The effect of bupivacaine skull block on the hemodynamic response to craniotomy. Anesth Analg. 1996 Dec;83(6):1256-61. doi: 10.1097/00000539-199612000-00022. PMID 8942596
- [Background] Jian M, Li X, Wang A, Zhang L, Han R, Gelb AW. Flurbiprofen and hypertension but not hydroxyethyl starch are associated with post-craniotomy intracranial haematoma requiring surgery. Br J Anaesth. 2014 Nov;113(5):832-9. doi: 10.1093/bja/aeu185. Epub 2014 Jun 25. PMID 24966149
- [Result] Osborn I, Sebeo J. "Scalp block" during craniotomy: a classic technique revisited. J Neurosurg Anesthesiol. 2010 Jul;22(3):187-94. doi: 10.1097/ANA.0b013e3181d48846. PMID 20479675
- See also: N. Narouze, S. (Ed.). (2014). Interventional Management of Head and Face Pain. — http://doi.org/10.1007/978-1-4614-8951-1
- See also: Tuchinda L, Somboonviboon W, Supbornsug K, Worathongchai S, Limutaitip S Asian biomedicine, 2010, 4(2), 243-251 — http://doi.org/10.2478/abm-2010-0031